CLINICAL TRIAL: NCT04956419
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Fluconazole Controlled, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of SHR8008 vs. Fluconazole in Subjects With Acute Vulvovaginal Candidiasis (VVC)
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR8008 vs. Fluconazole in Subjects With Acute Vulvovaginal Candidiasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8008-302
Record Dates: First submitted 2021-07-07; First posted 2021-07-09 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-07

CONDITIONS: Acute Vulvovaginal Candidiasis
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Fluconazole Controlled, Multicenter Phase III Clinical Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR8008 capsule
  Interventions: Drug: SHR8008 capsule
- Treatment group B (Active Comparator): Fluconazole capsule
  Interventions: Drug: Fluconazole capsule

INTERVENTIONS:
Drug: SHR8008 capsule — once daily for 2 days(Day 1 and Day 2),oral
  Arms: Treatment group A
Drug: Fluconazole capsule — once daily for 2 days(Every 72 hours) ,oral
  Arms: Treatment group B

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of SHR8008 vs. Fluconazole In Subjects with Acute vulvovaginal Candidiasis

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 and ≤75 years old;
2. Clinical diagnosis with VVC episodes at screening, signs and symptoms score of ≥ 7, with a documented positive potassium hydroxide (KOH) or Gram staining;
3. Subjects of childbearing potential must have a negative pregnancy test result at screening and agree to use highly effective contraceptive measures throughout the study;
4. Willing to sign the informed consent form to participate in this study.

Exclusion Criteria:

1. Have recurrent vulvovaginal candidiasis (RVVC) as defined by 4 or more confirmed VVC episodes in the past 12 months or history of RVVC;
2. Presence of concomitant vulvovaginitis caused by other pathogens;
3. History of cervical cancer, or "cervical intraepithelial neoplasia or malignancy" or "atypical squamous cells of undetermined significance (ASCUS)" as indicated by Pap test or other tests reported within 1 year before screening;
4. Moderate to severe hepatic and/or renal disorders;
5. Have received systemic or vulvovaginal antifungal drugs, antibacterials, antitrichomonal, CYP3A4 substrates or inducers or inhibitors, or vulvovaginal corticosteroids within 7 days prior to randomization;
6. Have received any estrogen replacement therapy or vaginal topical products within 7 days prior to randomization;
7. Have received systemic corticosteroid therapy within 30 days or systemic immunosuppressant therapy within 90 days prior to randomization;
8. Presence of significant laboratory abnormalities at screening;
9. QTc interval greater than 470 ms or other clinically significant ECG abnormalities at screening;
10. Have planned surgeries or other medical procedures that may impact compliance with the protocol;
11. Known history of hypersensitivity or intolerance to azole antifungal drugs;
12. Being in the menstrual period, pregnant, or lactating at screening, or planning to become pregnant during the study period;
13. History of narcotic or drug abuse or alcoholism within 6 months prior to screening;
14. Have participated in another clinical study and received the investigational drug containing active ingredient within 30 days prior to screening;
15. Other conditions unsuitable for participation in the study per investigator's judgment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2021-04-24 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with therapeutic cure | Day 28
  defined as absence of signs and symptoms of VVC plus negative culture of vaginal swabs for growth of Candida species

SECONDARY OUTCOMES:
The proportion of subjects therapeutic cure | Day 14
The proportion of subjects with clinical cure | Day 14 and Day 28
  defined as absence of signs and symptoms of VVC
The proportion of subjects with mycological cure | Day 14 and Day 28
  defined as negative culture of vaginal swabs for growth of Candida species
Changes from baseline in VVC signs and symptoms score | Day 14 and Day 28
The proportion of subjects receiving rescue therapy during the study | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China